CLINICAL TRIAL: NCT01469494
Title: A Randomized Clinical Trial Comparing Breast and Abdominal Related Morbidity of DIEP and SIEA Flaps
Brief Title: Breast and Abdominal Related Morbidity of DIEP and SIEA Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Keeping Abreast Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2011:120
Record Dates: First submitted 2011-10-23; First posted 2011-11-10 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2014-08

CONDITIONS: DIEP Flap Breast Reconstruction; SIEA Flap Breast Reconstruction
Keywords: DIEP flap; SIEA flap; breast reconstruction; objective isokinetic abdominal strength testing; fat necrosis; flap loss; seroma rate; abdominal wound breakdown; Breast-Q; abdominal wall outcome questionnaire
MeSH Terms: conditions — Fat Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DIEP flap group (Active Comparator): The standard of care for the patient population is the DIEP or SIEA flap breast reconstruction. Currently the single operating surgeon in the study will always try to perform a SIEA flap reconstruction. If the anatomy does not allow it he will convert to a DIEP flap. The majority of breast surgeons in North America will generally perform a DIEP flap initially. The proposed study does not alter the standard of care received.
  Interventions: Procedure: DIEP flap breast reconstruction
- SIEA flap group (Active Comparator): The standard of care for the patient population is the DIEP or SIEA flap breast reconstruction. Currently the single operating surgeon in the study will always try to perform a SIEA flap reconstruction. If the anatomy does not allow it he will convert to a DIEP flap. The majority of breast surgeons in North America will generally perform a DIEP flap initially. The proposed study does not alter the standard of care received.
  Interventions: Procedure: SIEA flap breast reconstruction

INTERVENTIONS:
Procedure: DIEP flap breast reconstruction — DIEP stands for deep inferior epigastric perforator. This is the name of the main blood vessel that runs through the abdominal tissue that will be used to reconstruct the breast. In DIEP flap reconstruction, only skin, fat, and blood vessels are removed from the lower belly (the abdomen between the waist and hips). No muscle is removed.
  Arms: DIEP flap group
Procedure: SIEA flap breast reconstruction — The SIEA flap is very similar to the DIEP flap procedure. Both techniques use the lower abdominal skin and fatty tissue to reconstruct a natural, soft breast following mastectomy.
  The main difference between the SIEA flap and the DIEP flap is the artery used to supply blood flow to the new breast. The SIEA blood vessels are found in the fatty tissue just below skin whereas the DIEP blood vessels run below and within the abdominal muscle (making the surgery more technically challenging). While the surgical preparation is slightly different, both procedures spare the abdominal muscle and only use the patient's skin and fat to reconstruct the breast.
  Arms: SIEA flap group

SUMMARY:
The Deep Inferior Epigastric Perforator flap (DIEP) is the current standard of care in breast reconstruction. The newer Superficial Inferior Epigastric Artery flap (SIEA) is felt to be an improvement as it does not damage the abdominal wall. The SIEA unfortunately has smaller vessels which put the flap at a higher risk of developing flap loss and fat necrosis. The uncertainty regarding the tradeoffs inherent in the choice of procedure has not been resolved. As such the investigators aim to perform a randomized single blinded trial to evaluate the abdominal and breast related morbidity associated with DIEP and SIEA flaps.

DETAILED DESCRIPTION:
A blinded, randomized, prospective clinical trial is being performed involving Manitoban women over 18 years undergoing unilateral or bilateral breast reconstruction. Women were originally randomized 50/50 to either the DIEP or SIEA group. Due to only about 60-70% of patients randomized to the SIEA group actually receiving the SIEA procedure, the weight of the randomization has now been changed to 70/30 (SIEA/DIEP) for the remainder of the study (approx. 40/110 recruited patients waiting for their OR). Objective isokinetic abdominal strength testing is being done pre-operatively and 3, 6 and 12 months post-operatively. A self-administered validated abdominal wall and breast outcome questionnaire (Breast-Q) is also given preoperatively and at 3 and 12 months postoperatively in . Secondary outcomes measured include: fat necrosis, abdominal wound breakdown, flap loss and seroma rate. Fat necrosis is detected using ultrasonography. Abdominal wound breakdown is measured using calipers. Seroma rates are tabulated and drainage volumes measured. Statistical analyses include a combination of parametric and non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* female subject older than 18
* with satisfactory abdominal tissue for DIEP and SIEA flap reconstruction
* fluent in English

Exclusion Criteria:

* reconstruction planned using latissimus dorsi flap, gluteal artery perforator flap or tissue expansion
* suffer from neurological back problems
* suffer form inguinal hernias

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in objective isokinetic abdominal strength | pre-operative (baseline), 3, 6 and 12 months post-operative
  Strength of the abdominal muscles and the back extensors is being objectively measured by isokinetic strength testing on an isokinetic dynamometer (Biodex System III with dual position back extension/flexion attachment). The abdominal strength testing is being performed pre-operatively and at 3, 6 and 12 months post-op. Objective measurements are used to address the strength of the rectus abdominus muscle and all data is collected by personnel at PanAn Clinic who have been trained in the required techniques. The technician performing the assessments is blinded to the type of breast reconstruction that has been performed.

SECONDARY OUTCOMES:
Breast-Q questionnaire | pre-operative (baseline) and 3 and 12 months post-operative
  self-administered and validated.
Fat Necrosis | 3 and 6 months post-operative
  Will be detected using ultrasonography. Ultrasound characteristics of fat necrosis are quite variable and reflect the degree of fibrosis. Assessment for fat necrosis will take place both 3 and 6 months post-operatively by another plastic surgeon who is therefore blinded to the procedure performed.
Seroma Rate and Drainage Volumes | 1 week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op
  Rates will be tabulated and drainage volumes will be measured during regular followup appointments with the care team (1 week post-op, 2 weeks post-op, 6-8 weeks post-op, 3 months post-op).
Flap Loss | 1 week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op
  Partial flap loss defined as tissue loss greater than 10 percent of the flap or fat necrosis greater than 5cm in diameter. Total flap loss will also be assessed. These assessments will be done during regular followup appointments with the care team (1 week post-op, 2 weeks post-op, 6-8 weeks post-op, 3 months post-op)
Abdominal Wound Breakdown | 1 week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op
  Defined as necrosis or wound dehiscence resulting in an open wound. Will be assessed with calipers. This will be assessed during regular followup appointments with the care team (1 week post-op, 2 weeks post-op, 6-8 weeks post-op, 3 months post-op)
Intra-Operative Outcomes: | Intra-operative
  Intra-operative data is also being collected with the intention of using it to identify any variables of the DIEP and SIEA procedures associated with the breast and abdominal outcomes being assessed in the study. The intra-operative data being collected includes whether or not the superficial inferior epigastric vessels are present in both treatment groups. If the vessels are present, it is recorded whether or not they are of sufficient calibre to support an SIEA flap. This information is to show how many patients enrolled would be candidates to receive the SIEA procedure had they not been randomized to a treatment group pre-operatively. The size of the SIEA/DIEA at the femoral artery/external iliac artery and the size of the SIEV/DIEV at the femoral vein/external iliac vein is also recorded, along with the size of the venous coupler used to anastomose the donor and recipient vein. Other intra-op. data is being collected as well.
Clinical Abdominal Examination | 1 week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op
  Patients are examined in the plastic surgery department both in the supine and upright positions for asymmetric positioning of the umbilicus, abdominal wall asymmetry, lower abdominal bulging, hernias and abdominal wound breakdown (post- operatively using calipers). Any pre-existing scars are also noted to see if this affects complication rates. This clinical examination is completed pre-operatively by the operating surgeon and during the regular follow-up appointments (1 week, 2 weeks, 6-8 weeks, 3 months post-op) by the head nurse, who has been instructed to do these assessments on every patient receiving DIEP or SIEA breast reconstruction. She therefore, does not know who is actually enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Blair R Peters, BSc, Principal Investigator — University of Manitoba Faculty of Medicine
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Selber JC, Fosnot J, Nelson J, Goldstein J, Bergey M, Sonnad S, Serletti JM. A prospective study comparing the functional impact of SIEA, DIEP, and muscle-sparing free TRAM flaps on the abdominal wall: Part II. Bilateral reconstruction. Plast Reconstr Surg. 2010 Nov;126(5):1438-1453. doi: 10.1097/PRS.0b013e3181ea42ed. PMID 21042100
- [Background] Selber JC, Nelson J, Fosnot J, Goldstein J, Bergey M, Sonnad SS, Serletti JM. A prospective study comparing the functional impact of SIEA, DIEP, and muscle-sparing free TRAM flaps on the abdominal wall: part I. unilateral reconstruction. Plast Reconstr Surg. 2010 Oct;126(4):1142-1153. doi: 10.1097/PRS.0b013e3181f02520. PMID 20885239
- [Background] Futter CM, Webster MH, Hagen S, Mitchell SL. A retrospective comparison of abdominal muscle strength following breast reconstruction with a free TRAM or DIEP flap. Br J Plast Surg. 2000 Oct;53(7):578-83. doi: 10.1054/bjps.2000.3427. PMID 11000074
- [Background] Blondeel N, Vanderstraeten GG, Monstrey SJ, Van Landuyt K, Tonnard P, Lysens R, Boeckx WD, Matton G. The donor site morbidity of free DIEP flaps and free TRAM flaps for breast reconstruction. Br J Plast Surg. 1997 Jul;50(5):322-30. doi: 10.1016/s0007-1226(97)90540-3. PMID 9245865
- [Background] Bonde CT, Lund H, Fridberg M, Danneskiold-Samsoe B, Elberg JJ. Abdominal strength after breast reconstruction using a free abdominal flap. J Plast Reconstr Aesthet Surg. 2007;60(5):519-23. doi: 10.1016/j.bjps.2006.07.003. Epub 2007 Jan 17. PMID 17399661